CLINICAL TRIAL: NCT02359877
Title: Open Label Study of Tolerability, Pharmacokinetics and Pharmacodynamics of BCD-054 (Pegylated Interferon Beta-1a), IM and SC, Compared to Rebif® and Avonex® in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biocad (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BCD-054-1
Record Dates: First submitted 2015-01-20; First posted 2015-02-10 (Estimated); Results first posted 2016-12-23 (Estimated); Last update posted 2017-04-10 (Actual); Status verified 2017-04

CONDITIONS: Healthy
Keywords: pegylated interferon beta; Volunteers
MeSH Terms: interventions — sampeginterferon beta-1a; Interferon beta-1a

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- BCD-054 (Experimental): Pegylated interferon beta 1a Single doses - 60 mcg, SC/IM Single doses - 120 mcg, SC/IM Single doses - 240 mcg, SC/IM Single doses - 360 mcg, SC/IM Multiple doses - 180 mcg, SC/IM
  Interventions: Drug: BCD-054
- Rebif (Active Comparator): interferon beta 1a 44 mcg, SC, 3 times a week for 2 weeks
  Interventions: Drug: Rebif
- Avonex (Active Comparator): interferon beta 1a 30 mcg, IM, once a week for 2 weeks
  Interventions: Drug: Avonex

INTERVENTIONS:
Drug: BCD-054
  Other Names: pegylated interferon beta 1a
  Arms: BCD-054
Drug: Rebif
  Other Names: interferon beta 1a
  Arms: Rebif
Drug: Avonex
  Other Names: interferon beta 1a
  Arms: Avonex

SUMMARY:
This is an international multicenter study of tolerability, pharmacokinetics and pharmacodynamics of drug product BCD-054 (CJSC BIOCAD, Russia), administrated intramuscular and subcutaneous, compared to Rebif® (Merck Serono S.p.A., Italy) and Avonex® (Biogen Idec Ltd, UK) in healthy volunteers. The study involves 2 stages - single ascending dose administration and multiple estimated therapeutic dose administration of BCD-054.

ELIGIBILITY:
InInclusion Criteria:

1. Written informed consent;
2. Male gender;
3. Age 18 - 45 years inclusive;
4. Body mass index (BMI) (18,5 - 24,99 kg/m2);
5. Healthy condition proven by the volunteer's history, global assessment and laboratory analysis results:

   * Absence in past medical history and at screening of clinically significant dysfunctions of circulatory, respiratory, nervous, hematopoietic, endocrine and digestive systems, liver and kidneys;
   * No history of cardiovascular diseases and diseases of the thyroid gland
   * Haematology and biochemistry tests, urinalysis and thyroid hormone analysis results are within normal limits according to standards of the study site. Screening laboratory analyses should be performed not more than 14 days before volunteer's inclusion in the study;
   * Hemodynamic parameters are within normal limits: systolic blood pressure - from 100 to 139 mmHg, diastolic blood pressure - from 60 to 90 mmHg, heart rate - from 50 to 90 bpm;
   * Absence of history of chronic infection (tuberculosis) and chronic inflammation;
   * Absence of HIV, hepatitis B and C virus, syphilis;
   * Absence of acute infections within 4 weeks before inclusion in the study;
   * Absence of psychiatric disorders and other conditions that can interfere with volunteer's ability to follow the study protocol, including depression;
   * Well-being (in volunteer's opinion) within 30 days before participation in the study;
6. Absence of history of systematic alcohol and drug abuse;
7. Ability of the volunteer, in investigator's opinion, to follow the study protocol procedures and requirements;
8. Willingness of volunteers and their sexual partners of childbearing potential to use reliable contraception methods starting from 2 weeks before inclusion into the study and until 4 weeks after receiving the last dose of the investigational products. This criterion is not applicable to patients who underwent surgical sterilization. Reliable contraceptive measures include one barrier method in combination with one of the following methods: spermicides, intrauterine device or oral contraceptives used by participant's partner;
9. Consent to avoid alcohol intake within 24 hours before and 8 days after each administration of the test or reference drugs;
10. Consent to avoid grapefruit juice (or other products containing grapefruit) intake within 72 hours before and 8 days after each administration of the study or reference drugs.

Exclusion Criteria:

1. Previous use of IFN-β1-containing medications at any time before inclusion;
2. History of serious allergic reactions (anaphylaxis or multiple allergy);
3. Known allergy or intolerance to interferons or any other components of study or reference drugs or pegylated proteins;
4. Major surgery within 30 days before screening;
5. Impossibility to install venous catheter for blood sampling (e.g. because of skin disorders at the sites of venipuncture);
6. Diseases or other conditions that can interfere with the investigational drugs pharmacokinetics (e.g. chronic liver, kidney, blood, circulatory system, lung or neuroendocrine diseases, including diabetes mellitus and others);
7. History of fever over 40°С
8. History of increase in aminotransferases (ALT, AST) > 2.5 × ULN
9. History of epileptic seizures;
10. Depression and/or suicidal ideas, suicide attempts in history
11. Regular oral or parenteral use of any medications including over-the-counter drugs, vitamins and nutritional additives within less than 2 weeks before inclusion in the study;
12. Intake of medications, including over-the-counter drugs and biologically active additives that can influence hemodynamics, liver function etc. (barbiturates, omeprazole, cimetidine etc.) within less than 30 days before inclusion in the study;
13. Intake of medications that influence immune status (cytokines and their inductors, glucocorticoids etc.) within less than 30 days before inclusion in the study;
14. Vaccination within 4 weeks prior to inclusion
15. Smoking more than 10 cigarettes per day;
16. Subjects who consume more than 10 units of alcohol per week or who have history of alcohol abuse or evidence of drug/chemical abuse (one unit of alcohol equals ½ l [500 ml] of beer, one glass [200 ml] of wine or l shot glass [50 ml] of spirits);
17. Donation of 450 ml and more of blood or plasma within 2 months before inclusion in the study;
18. Participation in other clinical studies within less than 1 month before inclusion in the study or simultaneous participation in another clinical study;
19. Previous participation in this study

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2014-07; Primary Completion 2015-10 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ivan Sardaryan, PhD, Principal Investigator — OOO BioEk
Locations (1):
- OOO "BioEk", Saint Petersburg, Russia

RESULTS

PARTICIPANT FLOW:
Groups:
- BCD-054 (Single Doses): Pegylated interferon beta 1a (BCD-054) Single doses - 60 mcg, IM/SC; or 120 mcg, IM/SC; or 240 mcg, IM/SC; or 360 mcg, IM/SC
- Rebif: interferon beta 1a (Rebif) 44 mcg, SC, 3 times a week for 2 weeks
- Avonex: interferon beta 1a (Avonex) 30 mcg, IM, once a week for 2 weeks
- BCD-054 (Multiple Dose): Pegylated interferon beta 1a (BCD-054) Multiple dose - 180 mcg, IM/SC, biweekly, 3 injections
Period: Overall Study
Arm/Group | BCD-054 (Single Doses) | Rebif | Avonex | BCD-054 (Multiple Dose)
Started | 34 | 6 | 6 | 14
Completed | 33 | 6 | 6 | 11
Not Completed | 1 | 0 | 0 | 3
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Presented baseline measures relate to all volunteers who participated in Stage 1.
Groups:
- BCD-054 (Multiple Doses): Pegylated interferon beta 1a (BCD-054) Multiple dose - 180 mcg, IM/SC, biweekly, 3 injections
- Total: Total of all reporting groups
Arm/Group | BCD-054 (Single Doses) | Rebif | Avonex | BCD-054 (Multiple Doses) | Total
Number analyzed (Participants) | 33 | 6 | 6 | 11 | 56
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 33 | 6 | 6 | 11 | 56
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 23 [21 to 26] | 23 [21 to 26] | 23 [21 to 26] | 21 [20 to 31] | 23 [21 to 26]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 33 | 6 | 6 | 11 | 56

OUTCOME MEASURES:

1. Primary Outcome: AUC (0-168); AUC (0-336); AUC (0-672); AUC (0-∞ ) of Interferon (IFN) Beta-1a
Description: Stage 1 primary outcome measure for pharmacokinetics analysis. Area under concentration-time curve (AUC) of interferon (IFN) beta-1a from the moment of drug administration up to 168, 336, 648 hours respectively
Time Frame: 0 to 168 hours; 0 to 336 hours; 0 to 672 hours respectively
Measure: Median (Inter-Quartile Range); unit: (pg/ml)*hour
Groups:
- BCD-054 - 60 mcg - SC: Pegylated interferon beta 1a (BCD-054) Single dose - 60 mcg, subcutaneously
- BCD-054 - 60 mcg - IM: Pegylated interferon beta 1a (BCD-054) Single dose - 60 mcg, intramuscular injection
- BCD-054 - 120 mcg - SC: Pegylated interferon beta 1a (BCD-054) Single dose - 120 mcg, subcutaneously
- BCD-054 - 120 mcg - IM: Pegylated interferon beta 1a (BCD-054) Single dose - 120 mcg, intramuscular injection
- BCD-054 - 240 mcg - SC: Pegylated interferon beta 1a (BCD-054) Single dose - 240 mcg, subcutaneously
- BCD-054 - 240 mcg - IM: Pegylated interferon beta 1a (BCD-054) Single dose - 240 mcg, intramuscular injection
- BCD-054 - 360 mcg - SC: Pegylated interferon beta 1a (BCD-054) Single dose - 360 mcg, subcutaneously
- BCD-054 - 360 mcg - IM: Pegylated interferon beta 1a (BCD-054) Single dose - 360 mcg, intramuscular injection
Arm/Group | BCD-054 - 60 mcg - SC | BCD-054 - 60 mcg - IM | BCD-054 - 120 mcg - SC | BCD-054 - 120 mcg - IM | BCD-054 - 240 mcg - SC | BCD-054 - 240 mcg - IM | BCD-054 - 360 mcg - SC | BCD-054 - 360 mcg - IM | Rebif | Avonex
Number analyzed (Participants) | 3 | 3 | 6 | 6 | 3 | 3 | 6 | 3 | 6 | 6
(pg/ml)*hour
  AUC (0-168) | 36682 [20348 to 132888] | 87085 [53718 to 133586] | 279477 [237578 to 309910] | 176866 [119715 to 191402] | 405395 [130963 to 835348] | 420038 [265413 to 692759] | 1052951 [534763 to 1195047] | 376277 [227428 to 522273] | 20423 [18115 to 22919] | 5995 [5139 to 7093]
  AUC (0-336) | 44569 [24305 to 175568] | 103624 [53718 to 162221] | 345510 [309323 to 439732] | 196189 [136976 to 215301] | 426025 [149813 to 931966] | 437275 [288706 to 737144] | 1457973 [554150 to 1625676] | 407273 [243598 to 564684] | 36866 [33072 to 51379] | 6964 [6006 to 8067]
  AUC (0-672) | 44569 [24305 to 185094] | 107471 [53718 to 175510] | 351768 [329256 to 457232] | 196189 [136976 to 215301] | 426025 [149813 to 938358] | 437275 [288706 to 737144] | 1554173 [563062 to 1849940] | 410751 [247529 to 569632] | 53715 [42627 to 78467] | 7544 [6645 to 8596]
  AUC (0-∞ ) | 44569 [24305 to 185094] | 107471 [53718 to 175510] | 351768 [329256 to 457232] | 196189 [136976 to 215301] | 426025 [149813 to 938358] | 437275 [288706 to 737144] | 1562327 [563063 to 1872683] | 410751 [247529 to 569632] | 54774 [43128 to 78872] | 7544 [6645 to 8707]

2. Primary Outcome: AUC(0-last); AUC (0-∞ ) BCD-054 of Interferon (IFN) Beta-1a - 180 mcg - SC, BCD-054 - 180 mcg - IM
Description: Stage 2 primary outcome measure for pharmacokinetics analysis. Area under concentration-time curve (AUC) of interferon (IFN) beta-1a from the moment of drug administration until last quantifiable concentration
Time Frame: 0 to 672 hours
Measure: Median (Inter-Quartile Range); unit: (pg/ml)*hour
Groups:
- BCD-054 - 180 mcg - SC; BCD-054 - 180 mcg - IM: Pegylated interferon beta 1a (BCD-054)
Arm/Group | BCD-054 - 180 mcg - SC | BCD-054 - 180 mcg - IM
Number analyzed (Participants) | 5 | 6
(pg/ml)*hour
  AUC(0-last) | 274888 [228924 to 450286] | 210626 [152236 to 383557]
  AUC (0-∞) | 316204 [245890 to 484802] | 218817 [152236 to 383557]

3. Primary Outcome: AUC (0-168); AUC (0-336); AUC (0-672);AUC (0-∞ ) of Neopterin
Description: Stage 1 primary outcome measure for pharmacodynamics analysis. Area under concentration-time curve (AUC) of neopterin from the moment of drug administration until 168, 336, 648 hours respectively
Time Frame: 0 to 168 hours; 0 to 336 hours; 0 to 672 hours respectively
Measure: Median (Inter-Quartile Range); unit: nmol/L*hour
Arm/Group | BCD-054 - 60 mcg - SC | BCD-054 - 60 mcg - IM | BCD-054 - 120 mcg - SC | BCD-054 - 120 mcg - IM | BCD-054 - 240 mcg - SC | BCD-054 - 240 mcg - IM | BCD-054 - 360 mcg - SC | BCD-054 - 360 mcg - IM | Rebif | Avonex
Number analyzed (Participants) | 3 | 3 | 6 | 6 | 3 | 3 | 6 | 3 | 6 | 6
nmol/L*hour
  AUC (0-168) | 36681 [20348 to 132887] | 87084 [53717 to 133585] | 279477 [237578 to 309909] | 176865 [119715 to 191401] | 405394 [130963 to 835348] | 420038 [265413 to 692758] | 1052951 [534763 to 1195047] | 376277 [227427 to 522273] | 20423 [18115 to 22918] | 5995 [5138 to 7092]
  AUC (0-336) | 44569 [24304 to 175568] | 103624 [53717 to 162221] | 345509 [309322 to 439731] | 196189 [136976 to 215301] | 426024 [149812 to 931965] | 437275 [288706 to 737144] | 1457972 [554150 to 1625676] | 407273 [243597 to 564684] | 36865 [33071 to 51379] | 6964 [6006 to 8067]
  AUC (0-672) | 44569 [24304 to 185093] | 107471 [53717 to 175510] | 351767 [329256 to 457231] | 196189 [136976 to 215301] | 426024 [149812 to 938358] | 437275 [288706 to 737144] | 1554173 [563062 to 1849939] | 410750 [247529 to 569632] | 53714 [42626 to 78466] | 7544 [6644 to 8596]
  AUC (0-∞ ) | 44569 [24304 to 185093] | 107471 [53717 to 175510] | 351767 [329256 to 457231] | 196189 [136976 to 215301] | 426024 [149812 to 938358] | 437275 [288706 to 737144] | 1562327 [563062 to 1872682] | 410750 [247529 to 569632] | 54774 [43127 to 78871] | 7544 [6644 to 8707]

4. Primary Outcome: AUC(0-∞), AUC(0-last) of Neopterin
Description: Stage 2 primary outcome measure for pharmacodynamics analysis. Area under concentration-time curve (AUC) of neopterin from the moment of drug administration until last quantifiable concentration
Time Frame: 0 to 672 hours
Measure: Median (Inter-Quartile Range); unit: (nmol/L)*hour
Arm/Group | BCD-054 - 180 mcg - SC | BCD-054 - 180 mcg - IM
Number analyzed (Participants) | 5 | 6
(nmol/L)*hour
  AUC(0-∞) | 3757 [3334 to 4655] | 3431 [2568 to 3614]
  AUC(0-last) | 3303 [3118 to 4487] | 3242 [2568 to 3612]

5. Primary Outcome: Adverse Event (AE) and Serious Adverse Event (SAE) Incidence
Description: Stage 1
Time Frame: 4 weeks
Measure: Number; unit: participants
Arm/Group | BCD-054 - 60 mcg - SC | BCD-054 - 60 mcg - IM | BCD-054 - 120 mcg - SC | BCD-054 - 120 mcg - IM | BCD-054 - 240 mcg - SC | BCD-054 - 240 mcg - IM | BCD-054 - 360 mcg - SC | BCD-054 - 360 mcg - IM | Rebif | Avonex
Number analyzed (Participants) | 3 | 3 | 6 | 6 | 3 | 3 | 6 | 3 | 6 | 6
participants
  Serious) Adverse Events | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Other (Not Including Serious) Adverse Events | 3 | 3 | 6 | 6 | 3 | 3 | 6 | 3 | 6 | 3
  Elevated erythrocyte sedimentation rate | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
  Leucopenia | 2 | 2 | 6 | 3 | 2 | 2 | 6 | 2 | 2 | 3
  Lymphopenia | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 1 | 0 | 0
  Monocytopenia | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Monocytosis | 1 | 2 | 1 | 2 | 0 | 1 | 0 | 2 | 0 | 1
  Neutropenia | 2 | 2 | 3 | 2 | 2 | 2 | 6 | 2 | 5 | 3
  Plasmatization of lymphocytes | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Trombocytopenia | 1 | 1 | 2 | 0 | 2 | 0 | 6 | 2 | 2 | 0
  Vacuolation of cytoplasm of monocytes | 3 | 3 | 0 | 3 | 0 | 0 | 0 | 1 | 0 | 0
  Fever | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0
  Flu-like syndrome | 1 | 1 | 4 | 6 | 3 | 3 | 4 | 2 | 4 | 1
  Elevated ALT | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0
  Elevated AST | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
  Elevated gamma glutamil transferrase | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Hyperemia of injection site | 1 | 0 | 3 | 0 | 1 | 0 | 4 | 0 | 1 | 0

6. Primary Outcome: Adverse Event (AE) and Serious Adverse Event (SAE) Incidence BCD-054 - 180 mcg - SC/IM
Description: Stage 2 BCD-054 - 180 mcg - SC/IM
Time Frame: 4 weeks
Measure: Number; unit: participants
Groups:
- BCD-054 - 180 mcg - SC: Pegylated interferon beta 1a (BCD-054) Single dose - 180 mcg, subcutaneously
- BCD-054 - 180 mcg - IM: Pegylated interferon beta 1a (BCD-054) Single dose - 180 mcg, intramuscular injection
Arm/Group | BCD-054 - 180 mcg - SC | BCD-054 - 180 mcg - IM
Number analyzed (Participants) | 8 | 6
participants
  Serious Adverse Events | 0 | 0
  Other (Not Including Serious) Adverse Events | 8 | 6
  Leucopenia | 4 | 6
  Neutropenia | 5 | 5
  Trombocytopenia | 1 | 3
  Flu-like syndrome | 7 | 4
  Elevated ALT | 3 | 2
  Elevated AST | 3 | 2
  Elevated creatinine | 0 | 1
  Hyperemia of injection site | 1 | 0

ADVERSE EVENTS:
Time Frame: 29 days after injection
Arm/Group | BCD-054 - 60 mcg - SC | BCD-054 - 60 mcg - IM | BCD-054 - 120 mcg - SC | BCD-054 - 120 mcg - IM | BCD-054 - 240 mcg - SC | BCD-054 - 240 mcg - IM | BCD-054 - 360 mcg - SC | BCD-054 - 360 mcg - IM | Rebif | Avonex | BCD-054 - 180 mcg - SC | BCD-054 - 180 mcg - IM
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/6 | 0/6 | 0/3 | 0/3 | 0/6 | 0/3 | 0/6 | 0/6 | 0/8 | 0/6
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 6/6 | 6/6 | 3/3 | 3/3 | 6/6 | 3/3 | 6/6 | 3/6 | 8/8 | 6/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BCD-054 - 60 mcg - SC (N=3) | BCD-054 - 60 mcg - IM (N=3) | BCD-054 - 120 mcg - SC (N=6) | BCD-054 - 120 mcg - IM (N=6) | BCD-054 - 240 mcg - SC (N=3) | BCD-054 - 240 mcg - IM (N=3) | BCD-054 - 360 mcg - SC (N=6) | BCD-054 - 360 mcg - IM (N=3) | Rebif (N=6) | Avonex (N=6) | BCD-054 - 180 mcg - SC (N=8) | BCD-054 - 180 mcg - IM (N=6)
Neutropenia (Blood and lymphatic system disorders) | 2 | 2 | 3 | 2 | 2 | 2 | 6 | 2 | 5 | 3 | 5 | 5
Monocytosis (Blood and lymphatic system disorders) | 1 | 2 | 1 | 2 | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 0
Vacuolation of cytoplasm of monocytes (Blood and lymphatic system disorders) | 3 | 3 | 0 | 3 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Leucopenia (Blood and lymphatic system disorders) | 2 | 2 | 6 | 3 | 2 | 2 | 6 | 2 | 2 | 3 | 4 | 6
Flu-like syndrome (General disorders) | 1 | 1 | 4 | 6 | 3 | 3 | 4 | 2 | 4 | 1 | 7 | 4
Hyperemia of injection site (Skin and subcutaneous tissue disorders) | 1 | 0 | 3 | 0 | 1 | 0 | 4 | 0 | 1 | 0 | 1 | 0
Trombocytopenia (Blood and lymphatic system disorders) | 1 | 1 | 2 | 0 | 2 | 0 | 6 | 2 | 2 | 0 | 1 | 3
Elevated erythrocyte sedimentation rate (Blood and lymphatic system disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Plasmatization of lymphocytes (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Elevated ALT (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 3 | 2
Elevated AST (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 3 | 2
Fever (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0
Monocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Elevated gamma glutamil transferrase (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 1 | 0 | 0 | 0 | 0
Elevated creatinine (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No